CLINICAL TRIAL: NCT03895125
Title: The Learning Effects of Attentional Strategy on Dual-task Walking in Patients With Parkinson's Disease: Behavioral Performance and Neural Plasticity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201812110RINC
Record Dates: First submitted 2019-03-13; First posted 2019-03-29 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease
Keywords: dual-task training; attention; Parkinson's disease; walking; EEG
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- [year1] PD group (Experimental)
  Interventions: Behavioral: [year1] dual-task training with task priority strategy
- [year1] healthy control group (Active Comparator)
  Interventions: Behavioral: [year1] dual-task training with task priority strategy
- [year2-3] freezer (Experimental)
  Interventions: Behavioral: [year2-3] dual-task training with internal and external focus
- [year2-3] non-freezer (Experimental)
  Interventions: Behavioral: [year2-3] dual-task training with internal and external focus

INTERVENTIONS:
Behavioral: [year1] dual-task training with task priority strategy — postural focus: focus mainly on postural performances while dual-tasking suprapostural focus: focus mainly on suprapostural performances while dual-tasking
  Arms: [year1] PD group; [year1] healthy control group
Behavioral: [year2-3] dual-task training with internal and external focus — internal focus: focus mainly on body movements external focus: focus mainly on object in the environment
  Arms: [year2-3] freezer; [year2-3] non-freezer

SUMMARY:
[year1]

1. To compare the effects of dual-task training with two different task priority instruction in people with Parkinson's disease and healthy controls on dual-task weight shifting performances.
2. Investigate the changes of brain activities and functional connectivity after dual-task training with different task priority instructions.

[year 2-3]

To investigate the learning effects of walking with internal/external focus on walking automaticity and brain plasticity in dual-task walking training for PD patients with/without freezing of gait.

DETAILED DESCRIPTION:
Postural-suprapostural task is defined as postural control takes place while another concurrent task is being performed, belonging to dual-task paradigms. Effective dual-task training is important to patients with Parkinson disease (PD), because they often lose balance and fall in dual-task conditions. Attentional strategy includes 1) task-priority between postural and suprapostural tasks and 2) internal and external focus for the postural task, which is the critical factor for both dual-task control and motor learning. However, the appropriateness of attentional strategy has not been investigated in dual-task training in patients with PD. Besides, there is lack of neural evidence of brain plasticity for previous studies about dual-task training in patients with PD. With the uses of EEG, EMG and behavioral measures, the purpose of this 3-year research project is to investigate the differences in performance quality and intrinsic neural mechanisms of dual-task training in PD, by adopting task-priority strategy and internal/external strategy during weight-shifting and walking. In the first year, the investigators will characterize task-priority effect (posture-priority vs. supraposture-priority) on dual-task training, with a special focus on modulation of brain plasticity and muscle activity patterns in weight-shifting posture for patients with PD. In the second and third years, the learning effects of walking internal/external focus on walking automaticity and brain plasticity will be investigated in dual-task walking training for PD patients with/without freezing of gait. Besides, the transfer effects of dual-task learning will be also investigated on medication "off" state. The present project is expected to have significant contributions not only to gain a better insight to neural correlates of dual-task training with different attentional strategies under weight-shifting and walking, but to optimize treatment strategy for PD patients with balance or dual-tasking disturbances.

ELIGIBILITY:
[year1]

Inclusion criteria:

1. For people with Parkinson's disease

   1. modified Hoehn & Yahr stage 2-3
   2. without dementia and able to follow instructions
2. For healthy controls

age and gender matched healthy subjects as control group

Exclusion criteria:

1. MMSE < 26
2. with other disease that may influence balance ability
3. with marked action and postural tremor

[year2-3] inclusion criteria:

1. idiopathic Parkinson's disease
2. modified Hoehn & Yahr stage 2-3
3. without marked action or postural tremor

exclusion criteria:

1. MMSE < 26
2. with other disease that may influence balance ability

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
postural performance | about 36 seconds for each trial for a total of 25 minutes
  measuring the amount of body weight shifting (unit: kg)
suprapostural performance | about 36 seconds for each trial for a total of 25 minutes
  measuring the rotation angle of box on the hand (unit: degree)
Walking speed | about 10-20 seconds for each trial
  collecting by using the GAITRite electronic walkway (CIR systems, Inc. ,USA) 24 inches(61cm) wide and 192 inches (488cm, 16ft) long, total 18,432 sensor (unit: m/s)
Cadence | about 10-20 seconds for each trial
  collecting by using the GAITRite (unit: step/s)
Gait symmetry | about 10-20 seconds for each trial
  collecting single leg supporting time of right and left leg by using the GAITRite

SECONDARY OUTCOMES:
electroencephalography (EEG) | about 36 seconds for each trial for a total of 25 minutes
  to collect the brain activity (unit: uV)
electromyography (EMG) | about 36 seconds for each trial for a total of 25 minutes
  to collect the muscle activity (unit: mV)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Ya Huang, Principal Investigator — School & Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan